CLINICAL TRIAL: NCT04046432
Title: Effects of Vigiis 101-LAB on Gut Health
Brief Title: Effects of Vigiis 101-LAB on a Healthy Populations' Gut Microflora, Peristalsis, Immunity, and Anti-oxidative Capacity
Acronym: Vigiis101
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SunWay Biotech Co., LTD. (Industry)
Collaborators: National Taiwan University Hospital (Other); Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: sunway 001
Record Dates: First submitted 2019-07-24; First posted 2019-08-06 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Gastrointestinal Microbiome
Keywords: gut microflora; immunity; anti-oxidative capacity; Lactobacillus paracasei subsp. paracasei NTU 101; probiotics

STUDY DESIGN:
Intervention Model Description: a randomized, double-blind, placebo-controlled clinical study
Who Masked: Participant
Masking Description: a randomized, double-blind, placebo-controlled clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vigiis 101-LAB (Experimental): The Vigiis 101-LAB mixed lactose, crystalline cellulose, and excipient were made into capsules (Vigiis 101-LAB capsule I) containing 5 billion bacteria per capsule for the gut flora clinical trial 1. The Vigiis 101-LAB mixed lactose, crystalline cellulose, and excipient were also mixed into capsules (Vigiis 101-LAB capsule II) containing 10 billion bacteria per capsule for clinical trial 2.
  Interventions: Dietary Supplement: Vigiis 101-LAB
- placebo (Placebo Comparator): Maltodextrin was used as a placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vigiis 101-LAB — examined the effects of the Vigiis 101-LAB capsules I or II (5 or 10 billion CFU/day)
  Arms: Vigiis 101-LAB
Dietary Supplement: Placebo — Maltodextrin was used as a placebo.
  Arms: placebo

SUMMARY:
Vigiis 101-LAB capsules I and II are produced from the fermentation of Lactobacillus paracasei subsp. paracasei NTU 101. Investigators have examined the effects of the Vigiis 101-LAB capsules I or II (5 or 10 billion CFU/day, respectively) on gut microflora in clinical trial 1, and on peristalsis, related immunity, and anti-oxidative capacity in clinical trial 2, during a 4-week randomized, double-blind, placebo-controlled, adaptive-design study.

DETAILED DESCRIPTION:
Detailed Description:

1.1 Lactobacillus paracasei subsp. paracasei NTU 101 strain (NTU 101) is a local Lactobacillus strain that was isolated and selected from the guts of newborns in Taiwan and shows good adaptability, gastric acid resistance, and bile salt resistance characteristics. This strain can survive for long periods in the human gut, inhibit the growth of harmful bacteria, and play multiple roles. Studies have shown that the NTU 101 strain, or its fermented products, contribute to several functions, namely: (1) improving the function of gut microflora by preventing harmful bacteria from colonizing the gut, thereby exerting protective effects; (2) regulating the immune system by stimulating cell activation and proliferation and increasing the secretion of cytokines and antibodies to enhance innate and acquired immune responses; (3) repairing damage to the gastric mucosa by inhibiting acute gastric mucosal injury caused by pylorus ligation and acidified alcohol, decreasing lipid peroxide concentrations in the blood and gastric mucosa, increasing the activity of superoxide dismutase, and promoting the synthesis of prostaglandin E2, which protects the mucosa; and (4) the improvement of gastrointestinal functions that contribute to alleviating metabolic abnormalities by improving gastrointestinal function and metabolism. This study is divided into two sections and focuses on Lactobacillus supplementation effects on healthy people using NTU 101. Investigators conducted clinical trials to assess the effects of the Vigiis 101-LAB capsule I on improving gastrointestinal function and regulating gut flora (clinical trial 1), and the Vigiis 101-LAB capsule II on the improvement of peristalsis, immunity, and anti-oxidative capacity (clinical trial 2).

1.2 Materials The strain used in the current study was L. paracasei subsp. paracasei NTU 101 (lyophilized powdered, Vigiis 101-LAB; probiotic powder from SunWay Biotech Co., Ltd., Taipei, Taiwan). The Vigiis 101-LAB mixed lactose, crystalline cellulose, and excipient were made into capsules (Vigiis 101-LAB capsule I) containing 5 billion bacteria per capsule for the gut flora clinical trial 1. The Vigiis 101-LAB mixed lactose, crystalline cellulose, and excipient were also mixed into capsules (Vigiis 101-LAB capsule II) containing 10 billion bacteria per capsule for clinical trial 2 on peristalsis, immunity, and anti-oxidative capacity. Maltodextrin was used as a placebo.

1.3 Randomized, double-blind clinical criteria of effects of Vigiis 101-LAB capsule I on gut flora (clinical trial 1) Vigiis 101-LAB capsule I was administered orally once per day, one capsule each time. The entire study took 4 weeks, and subjects were prohibited from eating fermented food products, such as miso, kimchi, fermented dairy products, oligosaccharide-containing foods, and lactic acid bacteria-containing products. Subjects also avoided consuming excessive gas-producing foods (such as soybeans and sweet potatoes) during their daily meals and avoided foods that can cause abdominal distension or promote peristalsis (such as lactic acid beverages and oligosaccharide-containing beverages). After the trial started, subjects recorded their daily number of bowel movements and completed relevant questionnaires at weeks 0, 2, and 4. The subjects visited the doctor once every 2 weeks for monitoring gastrointestinal function and physiological characteristics. At weeks 0, 1, 2, 3, and 4, fecal samples from the subjects were collected and put into bottles containing an anaerobic diluent and shaken to uniformly mix the feces and diluent.

1.4 Randomized, double-blind clinical criteria for evaluating effects of Vigiis 101-LAB capsule II on peristalsis, immunity, and anti-oxidative capacity (clinical trial 2) Clinical trial 2 was conducted from March 2017 to April 2018 at the Chung Shan Medical University after acquiring approval from the IRB of the Taichung Chung Shan Medical University Hospital (IRB proof document CHMUH No: CS17018), and all subjects signed an informed consent form. Vigiis 101-LAB capsule II was administered orally once per day, one capsule each time. Every day, the diet of the subjects was recorded in detail from the pre-stability to post-stability period.

1.5 Outcome measurements Fecal moisture content and pH value testing. Anthropometric measurements included the body height (BH), body weight (BW), blood pressure (BP), midarm circumference (MAC), triceps skinfold (TSF), waist circumference (WC), and rump circumference (RC) and heart rate (HR) were measured. The body mass index (= BW/BH2, kg/m2) of the subjects was calculated after measuring their BH and BW. For blood pressure measurements, the systolic blood pressure (SBP) and diastolic blood pressure (DBP) of the right arm were measured. MAC was measured using the same pair of calipers by the same trained staff member. Biochemical tests of the fasting blood samples were collected at weeks 0, 4, and 6. The test items included blood biochemistry tests, plasma antioxidant activity (Trolox equivalent antioxidant capacity, TEAC), thiobarbituric acid reactive substances (TBARS), glutathione levels (GSH), glutathione peroxidase (GSH Px), glutathione reductase (GSH Rd), full blood count, and blood electrolytes. Blood biochemical tests were carried out in the laboratory.

1.6. Statistical analysis Data are expressed as the mean ± standard deviation (SD). The statistical significance of the biochemical analyses was determined by one-way analysis of variance (ANOVA) using the general linear model procedure of the statistical product and service solutions software (SPSS Institute, Inc., Chicago, IL, USA). This was followed by ANOVA with a paired t-test to evaluate the difference before and after sample and placebo administration, while the Student t-test was used to compare the difference between test and placebo groups (P ≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≧ 20 years and ≦ 65 years.
* Subjects with normal weight (body mass index: 18.5-24).
* Subjects with no gastrointestinal diseases or on medication.

Exclusion Criteria:

* Pregnant or lactating women.
* Subjects who are allergic to Lactobacillus.
* Subjects with chronic gastrointestinal diseases.
* Subjects who previously underwent gastrectomy or gastric bypass.
* Subjects with liver, kidney, or heart disease, alcoholism, or uncontrolled diabetes.
* Subjects who developed stroke, psychiatric diseases, or depression within the last 1 year.
* Subjects being administered drugs that can regulate gastrointestinal function, functional foods, bacteriostatic drugs or supplements, antibiotics, antioxidants, or other unknown drugs within the last 2 weeks.
* Patients who did not fulfill the inclusion criteria, did not administer the test product according to regulations, whose efficacy could not be determined, or who had incomplete data that affect efficacy or safety assessment.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Gut Microflora | 4 week
  Outcome measurements:
  Analysis of correlation between stool frequency and gut microbiota change of the gut microbiome will be calculated at 4 week in comparison with admission.
Peristalsis intestine | 6 week
  Analysis of correlation between chyme passage time through the gut at 4 and 6 week in comparison with admission.

CONTACTS AND LOCATIONS:
Overall Officials: Tsong Ming Lu, MD, Principal Investigator; Jyh Ming Liou, MD.,PHD, Study Director
Locations (1):
- Division of Gastroenterology and Hepatology, Department of Internal Medicine, National Taiwan University Hospital, National Taiwan University College of Medicine, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Effects of Vigiis 101-LAB capsule I on improving gut microflora was examined Effects of Vigiis 101-LAB capsule II on improving gut peristalsis was examined Vigiis 101-LAB capsule I increased Bifidobacterium spp. and Lactobacillus spp. counts Vigiis 101-LAB capsule II improved gut motility and decreased food transiting time Vigiis 101-LAB capsule II increased IgG, IgM, and antioxidant activity
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication.
Access Criteria: 醫療/護理 Medicine / Nursing
  Medical Doctor Healthcare / Medical Management Medical Technician Pharmacist Nurse / Nursing Personnel Clinical Coodinator Clinical Researcher

REFERENCES:
- [Result] Agace WW, McCoy KD. Regionalized Development and Maintenance of the Intestinal Adaptive Immune Landscape. Immunity. 2017 Apr 18;46(4):532-548. doi: 10.1016/j.immuni.2017.04.004. PMID 28423335
- [Result] Arnao MB, Cano A, Hernandez-Ruiz J, Garcia-Canovas F, Acosta M. Inhibition by L-ascorbic acid and other antioxidants of the 2.2'-azino-bis(3-ethylbenzthiazoline-6-sulfonic acid) oxidation catalyzed by peroxidase: a new approach for determining total antioxidant status of foods. Anal Biochem. 1996 May 1;236(2):255-61. doi: 10.1006/abio.1996.0164. PMID 8660502
- [Result] Atarashi K, Tanoue T, Shima T, Imaoka A, Kuwahara T, Momose Y, Cheng G, Yamasaki S, Saito T, Ohba Y, Taniguchi T, Takeda K, Hori S, Ivanov II, Umesaki Y, Itoh K, Honda K. Induction of colonic regulatory T cells by indigenous Clostridium species. Science. 2011 Jan 21;331(6015):337-41. doi: 10.1126/science.1198469. Epub 2010 Dec 23. PMID 21205640
- [Result] Belkaid Y, Hand TW. Role of the microbiota in immunity and inflammation. Cell. 2014 Mar 27;157(1):121-41. doi: 10.1016/j.cell.2014.03.011. PMID 24679531
- [Result] Belkaid Y, Harrison OJ. Homeostatic Immunity and the Microbiota. Immunity. 2017 Apr 18;46(4):562-576. doi: 10.1016/j.immuni.2017.04.008. PMID 28423337
- [Result] Bengmark S. Gut microbiota, immune development and function. Pharmacol Res. 2013 Mar;69(1):87-113. doi: 10.1016/j.phrs.2012.09.002. Epub 2012 Sep 16. PMID 22989504
- [Result] Bridgman SL, Azad MB, Field CJ, Haqq AM, Becker AB, Mandhane PJ, Subbarao P, Turvey SE, Sears MR, Scott JA, Wishart DS, Kozyrskyj AL; CHILD Study Investigators. Fecal Short-Chain Fatty Acid Variations by Breastfeeding Status in Infants at 4 Months: Differences in Relative versus Absolute Concentrations. Front Nutr. 2017 Apr 10;4:11. doi: 10.3389/fnut.2017.00011. eCollection 2017. PMID 28443284
- [Result] Chen T, Isomaki P, Rimpilainen M, Toivanen P. Human cytokine responses induced by gram-positive cell walls of normal intestinal microbiota. Clin Exp Immunol. 1999 Nov;118(2):261-7. doi: 10.1046/j.1365-2249.1999.01047.x. PMID 10540188
- [Result] Chiang SS, Pan TM. Antiosteoporotic effects of Lactobacillus -fermented soy skim milk on bone mineral density and the microstructure of femoral bone in ovariectomized mice. J Agric Food Chem. 2011 Jul 27;59(14):7734-42. doi: 10.1021/jf2013716. Epub 2011 Jun 21. PMID 21668014
- [Result] Chiang SS, Liu CF, Ku TW, Mau JL, Lin HT, Pan TM. Use of murine models to detect the allergenicity of genetically modified Lactococcus lactis NZ9000/pNZPNK. J Agric Food Chem. 2011 Apr 27;59(8):3876-83. doi: 10.1021/jf104656m. Epub 2011 Mar 29. PMID 21410287
- [Result] Chiu CH, Lu TY, Tseng YY, Pan TM. The effects of Lactobacillus-fermented milk on lipid metabolism in hamsters fed on high-cholesterol diet. Appl Microbiol Biotechnol. 2006 Jun;71(2):238-45. doi: 10.1007/s00253-005-0145-0. Epub 2005 Sep 20. PMID 16172889
- [Result] Landi M. Commentary to: "Improving the thiobarbituric acid-reactive-substances assay for estimating lipid peroxidation in plant tissues containing anthocyanin and other interfering compounds" by Hodges et al., Planta (1999) 207:604-611. Planta. 2017 Jun;245(6):1067. doi: 10.1007/s00425-017-2699-3. Epub 2017 Apr 29. No abstract available. PMID 28456836
- [Result] Hooper LV, Littman DR, Macpherson AJ. Interactions between the microbiota and the immune system. Science. 2012 Jun 8;336(6086):1268-73. doi: 10.1126/science.1223490. Epub 2012 Jun 6. PMID 22674334
- [Result] Kao L, Liu TH, Tsai TY, Pan TM. Beneficial effects of the commercial lactic acid bacteria product, Vigiis 101, on gastric mucosa and intestinal bacterial flora in rats. J Microbiol Immunol Infect. 2020 Apr;53(2):266-273. doi: 10.1016/j.jmii.2018.06.002. Epub 2018 Jun 23. PMID 29970350
- [Result] Kamada N, Seo SU, Chen GY, Nunez G. Role of the gut microbiota in immunity and inflammatory disease. Nat Rev Immunol. 2013 May;13(5):321-35. doi: 10.1038/nri3430. PMID 23618829
- [Result] Kechagia M, Basoulis D, Konstantopoulou S, Dimitriadi D, Gyftopoulou K, Skarmoutsou N, Fakiri EM. Health benefits of probiotics: a review. ISRN Nutr. 2013 Jan 2;2013:481651. doi: 10.5402/2013/481651. eCollection 2013. PMID 24959545
- [Result] Kleniewska P, Hoffmann A, Pniewska E, Pawliczak R. The Influence of Probiotic Lactobacillus casei in Combination with Prebiotic Inulin on the Antioxidant Capacity of Human Plasma. Oxid Med Cell Longev. 2016;2016:1340903. doi: 10.1155/2016/1340903. Epub 2016 Mar 14. PMID 27066188
- [Result] Kopp-Hoolihan L. Prophylactic and therapeutic uses of probiotics: a review. J Am Diet Assoc. 2001 Feb;101(2):229-38; quiz 239-41. doi: 10.1016/S0002-8223(01)00060-8. PMID 11271697
- [Result] Krasowska A, Sigler K. How microorganisms use hydrophobicity and what does this mean for human needs? Front Cell Infect Microbiol. 2014 Aug 19;4:112. doi: 10.3389/fcimb.2014.00112. eCollection 2014. PMID 25191645
- [Result] Lee N, Kim WU. Microbiota in T-cell homeostasis and inflammatory diseases. Exp Mol Med. 2017 May 26;49(5):e340. doi: 10.1038/emm.2017.36. PMID 28546563
- [Result] Lei E, Vacy K, Boon WC. Fatty acids and their therapeutic potential in neurological disorders. Neurochem Int. 2016 May;95:75-84. doi: 10.1016/j.neuint.2016.02.014. Epub 2016 Mar 3. PMID 26939763
- [Result] Lin FM, Chiu CH, Pan TM. Fermentation of a milk-soymilk and Lycium chinense Miller mixture using a new isolate of Lactobacillus paracasei subsp. paracasei NTU101 and Bifidobacterium longum. J Ind Microbiol Biotechnol. 2004 Dec;31(12):559-64. doi: 10.1007/s10295-004-0184-z. Epub 2004 Nov 18. PMID 15662546
- [Result] Liu CF, Hu CL, Chiang SS, Tseng KC, Yu RC, Pan TM. Beneficial preventive effects of gastric mucosal lesion for soy-skim milk fermented by lactic acid bacteria. J Agric Food Chem. 2009 May 27;57(10):4433-8. doi: 10.1021/jf900465c. Epub 2009 Apr 9. PMID 19358530
- [Result] Liu CF, Tung YT, Wu CL, Lee BH, Hsu WH, Pan TM. Antihypertensive effects of Lactobacillus-fermented milk orally administered to spontaneously hypertensive rats. J Agric Food Chem. 2011 May 11;59(9):4537-43. doi: 10.1021/jf104985v. Epub 2011 Apr 4. PMID 21446645
- [Result] Lobo V, Patil A, Phatak A, Chandra N. Free radicals, antioxidants and functional foods: Impact on human health. Pharmacogn Rev. 2010 Jul;4(8):118-26. doi: 10.4103/0973-7847.70902. PMID 22228951
- [Result] Miller NJ, Sampson J, Candeias LP, Bramley PM, Rice-Evans CA. Antioxidant activities of carotenes and xanthophylls. FEBS Lett. 1996 Apr 22;384(3):240-2. doi: 10.1016/0014-5793(96)00323-7. PMID 8617362
- [Result] Naidu AS, Bidlack WR, Clemens RA. Probiotic spectra of lactic acid bacteria (LAB). Crit Rev Food Sci Nutr. 1999 Jan;39(1):13-126. doi: 10.1080/10408699991279187. PMID 10028126
- [Result] Orrhage K, Sillerstrom E, Gustafsson JA, Nord CE, Rafter J. Binding of mutagenic heterocyclic amines by intestinal and lactic acid bacteria. Mutat Res. 1994 Dec 1;311(2):239-48. doi: 10.1016/0027-5107(94)90182-1. PMID 7526189
- [Result] Ouwehand AC, Isolauri E, Kirjavainen PV, Tolkko S, Salminen SJ. The mucus binding of Bifidobacterium lactis Bb12 is enhanced in the presence of Lactobacillus GG and Lact. delbrueckii subsp. bulgaricus. Lett Appl Microbiol. 2000 Jan;30(1):10-3. doi: 10.1046/j.1472-765x.2000.00590.x. PMID 10728552
- [Result] Ouwehand AC, Salminen S, Isolauri E. Probiotics: an overview of beneficial effects. Antonie Van Leeuwenhoek. 2002 Aug;82(1-4):279-89. PMID 12369194
- [Result] Pant N, Marcotte H, Brussow H, Svensson L, Hammarstrom L. Effective prophylaxis against rotavirus diarrhea using a combination of Lactobacillus rhamnosus GG and antibodies. BMC Microbiol. 2007 Sep 27;7:86. doi: 10.1186/1471-2180-7-86. PMID 17900343
- [Result] Perdigon G, Vintini E, Alvarez S, Medina M, Medici M. Study of the possible mechanisms involved in the mucosal immune system activation by lactic acid bacteria. J Dairy Sci. 1999 Jun;82(6):1108-14. doi: 10.3168/jds.S0022-0302(99)75333-6. PMID 10386296
- [Result] Pool-Zobel BL, Neudecker C, Domizlaff I, Ji S, Schillinger U, Rumney C, Moretti M, Vilarini I, Scassellati-Sforzolini R, Rowland I. Lactobacillus- and bifidobacterium-mediated antigenotoxicity in the colon of rats. Nutr Cancer. 1996;26(3):365-80. doi: 10.1080/01635589609514492. PMID 8910918
- [Result] Rafter J. The effects of probiotics on colon cancer development. Nutr Res Rev. 2004 Dec;17(2):277-84. doi: 10.1079/NRR200484. PMID 19079931
- [Result] Saavedra JM, Bauman NA, Oung I, Perman JA, Yolken RH. Feeding of Bifidobacterium bifidum and Streptococcus thermophilus to infants in hospital for prevention of diarrhoea and shedding of rotavirus. Lancet. 1994 Oct 15;344(8929):1046-9. doi: 10.1016/s0140-6736(94)91708-6. PMID 7934445
- [Result] Schuijt TJ, van der Poll T, de Vos WM, Wiersinga WJ. The intestinal microbiota and host immune interactions in the critically ill. Trends Microbiol. 2013 May;21(5):221-9. doi: 10.1016/j.tim.2013.02.001. Epub 2013 Feb 28. PMID 23454077
- [Result] Sekine K, Toida T, Saito M, Kuboyama M, Kawashima T, Hashimoto Y. A new morphologically characterized cell wall preparation (whole peptidoglycan) from Bifidobacterium infantis with a higher efficacy on the regression of an established tumor in mice. Cancer Res. 1985 Mar;45(3):1300-7. PMID 3971375
- [Result] Sheng Y, Yang X, Lian Y, Zhang B, He X, Xu W, Huang K. Characterization of a cadmium resistance Lactococcus lactis subsp. lactis strain by antioxidant assays and proteome profiles methods. Environ Toxicol Pharmacol. 2016 Sep;46:286-291. doi: 10.1016/j.etap.2016.08.008. Epub 2016 Aug 6. PMID 27522548
- [Result] Smith PM, Howitt MR, Panikov N, Michaud M, Gallini CA, Bohlooly-Y M, Glickman JN, Garrett WS. The microbial metabolites, short-chain fatty acids, regulate colonic Treg cell homeostasis. Science. 2013 Aug 2;341(6145):569-73. doi: 10.1126/science.1241165. Epub 2013 Jul 4. PMID 23828891
- [Result] Stecher B. The Roles of Inflammation, Nutrient Availability and the Commensal Microbiota in Enteric Pathogen Infection. Microbiol Spectr. 2015 Jun;3(3). doi: 10.1128/microbiolspec.MBP-0008-2014. PMID 26185088
- [Result] Sun Y, O'Riordan MX. Regulation of bacterial pathogenesis by intestinal short-chain Fatty acids. Adv Appl Microbiol. 2013;85:93-118. doi: 10.1016/B978-0-12-407672-3.00003-4. PMID 23942149
- [Result] Thursby E, Juge N. Introduction to the human gut microbiota. Biochem J. 2017 May 16;474(11):1823-1836. doi: 10.1042/BCJ20160510. PMID 28512250
- [Result] Tomkovich S, Jobin C. Microbiota and host immune responses: a love-hate relationship. Immunology. 2016 Jan;147(1):1-10. doi: 10.1111/imm.12538. Epub 2015 Nov 2. PMID 26439191
- [Result] Tsai TY, Chu LH, Lee CL, Pan TM. Atherosclerosis-preventing activity of lactic acid bacteria-fermented milk-soymilk supplemented with Momordica charantia. J Agric Food Chem. 2009 Mar 11;57(5):2065-71. doi: 10.1021/jf802936c. PMID 19216552
- [Result] Tsai YT, Cheng PC, Pan TM. Immunomodulating activity of Lactobacillus paracasei subsp. paracasei NTU 101 in enterohemorrhagic Escherichia coli O157H7-infected mice. J Agric Food Chem. 2010 Nov 10;58(21):11265-72. doi: 10.1021/jf103011z. Epub 2010 Oct 13. PMID 20942489
- [Result] Tsai YT, Cheng PC, Fan CK, Pan TM. Time-dependent persistence of enhanced immune response by a potential probiotic strain Lactobacillus paracasei subsp. paracasei NTU 101. Int J Food Microbiol. 2008 Dec 10;128(2):219-25. doi: 10.1016/j.ijfoodmicro.2008.08.009. Epub 2008 Aug 26. PMID 18809220
- [Result] Tuson HH, Weibel DB. Bacteria-surface interactions. Soft Matter. 2013 May 14;9(18):4368-4380. doi: 10.1039/C3SM27705D. PMID 23930134
- [Result] Van de Water J, Keen CL, Gershwin ME. The influence of chronic yogurt consumption on immunity. J Nutr. 1999 Jul;129(7 Suppl):1492S-5S. doi: 10.1093/jn/129.7.1492S. PMID 10395628
- [Result] Yu X, Li S, Yang D, Qiu L, Wu Y, Wang D, Shah NP, Xu F, Wei H. A novel strain of Lactobacillus mucosae isolated from a Gaotian villager improves in vitro and in vivo antioxidant as well as biological properties in D-galactose-induced aging mice. J Dairy Sci. 2016 Feb;99(2):903-914. doi: 10.3168/jds.2015-10265. Epub 2015 Dec 17. PMID 26709186